CLINICAL TRIAL: NCT06222424
Title: Emergency Medicine Pharmacist Prescriptive Authority for Resolution of Outpatient Prescription Issues: a Descriptive Study
Brief Title: Emergency Medicine Pharmacist Prescriptive Authority for Resolution of Outpatient Prescription Issues
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 045.PHA.2023.C
Record Dates: First submitted 2024-01-16; First posted 2024-01-24 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-10

CONDITIONS: Outpatient Prescription Issues

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients at MCMC who had a prescription sent by an EMP between November 1, 2021 and June 30, 2023 (Other): Evaluation of utility will involve describing all EMP-written prescriptions pursuant to resolution of prescription issues realized after discharge.
  Interventions: Other: outpatient prescription issues

INTERVENTIONS:
Other: outpatient prescription issues — Evaluation of utility will involve describing all Emergency Medicine Pharmacist (EMP)-written prescriptions pursuant to resolution of prescription issues realized after discharge

SUMMARY:
The study aims to document the utility of Methodist Charlton Medical Center (MCMC's)Emergency Medicine Pharmacist (EMP) Collaborative Practice Agreement (CPA )utilization for the resolution of outpatient prescription issues. Evaluation of utility will involve describing all EMP-written prescriptions pursuant to resolution of prescription issues realized after discharge.

DETAILED DESCRIPTION:
Use of an EMP CPA, which allows for broad prescriptive authority, will assist Emergency Department (ED )workflow by preventing a significant volume of new prescriptions needing to be sent by physician and mid-level providers. Will improve rates of ED re-visits. In addition, this Collaborative Practice Agreement (CPA) will not be associated with a large volume of new prescription errors.

ELIGIBILITY:
Inclusion Criteria:

* Patients at MCMC who had a prescription sent by an EMP between November 1, 2021 and June 30, 2023 and a progress note and documenting the reason for the call and action taken by the EMP.

Exclusion Criteria:

* CPA actions were misclassified as discharge prescription issue resolutions.
* Patients with prescriptions pursuant to late culture review, formulation changes not requiring a new prescription, prescription transfers to another pharmacy, or simple retransmission of prescriptions.
* Patients documented to have left the ED against medical advice.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of prescriptions and medication types sent to outpatient pharmacies | 2 years
  Number of prescriptions and medication types sent to outpatient pharmacies by EMPs pursuant to outpatient prescription issue resolution.

SECONDARY OUTCOMES:
Number of patients returning with complaint or diagnosis related to EMP generated prescriptions | 2 years
  Proportion of patients returning with a complaint or diagnosis related to index EMP-generated prescriptions at three and six-month time points

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Burnham, Pharm.D., Principal Investigator — Methodist Health System
Locations (1):
- Clinical Research Institute at Methodist Health System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No